CLINICAL TRIAL: NCT04743726
Title: Research on the Physiological Characteristics of the Gastrointestinal Tract in Chinese Volunteers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dongyang Liu (Other)
Responsible Party: Sponsor-Investigator, Dongyang Liu, Vice director of Drug Clinical Trial Center, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: CPPO-PKMS-01
Record Dates: First submitted 2021-01-27; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Endoscopy, Gastrointestinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Days
Biospecimen Retention: Samples With DNA — Retention the samples, including gastrointestinal mucosa tissue, gastric juice, saliva, feces and blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopy: Chinese volunteers who are scheduling for gastro-colonoscopy

SUMMARY:
The dissolution and absorption of oral drugs in the gastrointestinal tract is a complex process, which is affected by physiological factors such as transporters, metabolic enzymes, gene phenotypes, gastrointestinal diseases, intestinal flora and so on. Therefore, the investigators are planning to collect gastrointestinal mucosa tissues, gastric juice, saliva , feces and blood samples to investigate (1) the activity and abundance of metabolism enzymes/transports in different section of gastrointestinal tract, (2) the composition and physicochemical properties of gastric juice; (3) the distribution and abundance of bacterial in gastrointestinal mucosa, saliva, gastric juice and feces; (4) the composition and content of bile acid in gastrointestinal mucosa, gastric juice and plasma in Chinese volunteers who planning to undergo digestive endoscopy.

DETAILED DESCRIPTION:
This is a single-center, open-labelled study. Twenty four Chinese adult volunteers who schedule for gastrointestinal endoscopy will be enrolled and will be not allowed to take products containing grapefruit, fruit juice, tea, coffee, wine and other foods or drinks containing caffeine, xanthine and alcohols at least 14 days before the gastrointestinal endoscopes. In addition, smoking is also prohibited. Screen will be performed any day between 3 and 14 days prior to the gastrointestinal endoscopes. Feces, saliva and 4 ml whole blood samples will be collected from these participants 3 days before gastrointestinal endoscopes for the detection of bacterial diversity, metabolic enzymes, transporter-related genotypes and bile acids. Afterwards, participants will undergo painless gastroscopy. Meanwhile, gastric juice, mucosal tissue from stomach, duodenum, jejunum, ileum, colon will be collected. The total number of mucosal tissue no more than 10.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese volunteers who are planning to undergo digestive endoscopy;
2. Volunteers who have a full understanding of the content, process and possible adverse reactions of the study and have signed an informed consent form before the clinical trial;
3. Volunteers who are able to complete the clinical trial according to the protocol;
4. Male and female volunteers between the ages of 18 and 60 (including both ends) on the date of signing the consent form;
5. Female volunteers are non-pregnant or non-lactating women, and will live asexually after enrollment until the end of the trial;
6. Male volunteers weigh no less than 50 kg, female volunteers weigh no less than 45 kg, and the body mass index (BMI) of male and female volunteers within the range of 19.0-26.0 kg/m2 (including cut-off values);
7. The comprehensive physical examination, routine laboratory examinations are normal or abnormal, but the investigator judges that there is no clinical significance;
8. Volunteers who are able to abstain from alcohol, coffee, non-prescription drugs or prescription drugs, and no food and beverages related to grapefruit within 14 days before the start of the test until the end of the test;
9. Volunteers have no history of smoking

Exclusion Criteria:

1. Volunteers who disagree with "No food or beverages containing caffeine, xanthine and alcohols such as grapefruit-containing products, juice, tea, coffee, wine, etc., 14 days before endoscope", "No smoking 14 days before endoscope";
2. Volunteers who do not comply with the relevant regulations about endoscope;
3. Volunteers with endoscope contraindications;
4. Volunteers with HCV, HIV, HBsAg and/or syphilis positive antibody;
5. Volunteers with allergic physique;
6. Volunteers with needlesickness, blood phobia, difficult in collecting blood and in tolerating local anesthesia;
7. Females who are pregnant, breastfeeding, or taking birth control pills for less than 3 months;
8. Volunteers have bleeding disorders, or therapeutic anticoagulation (warfarin, aspirin, clopidogrel, traditional Chinese medicine, etc.), or anesthesia dependence or alcohol dependence;
9. Volunteers have the smoking history, alcoholism history, alcohol screening positive, drug screening positive, history of drug abuse in the past five years or administration drugs in the three months prior to the trial;
10. Alcoholics (14 units of alcohol consumed per week: 1 unit = 285 mL beer, or 25 mL spirits, or 100 mL wine) and volunteers who cannot prohibition from the time of enrollment to the end of the study;
11. Volunteers who have a history of gastrointestinal disease with a definite severity or have diseases that have been considered unsuitable for participating in this study by researchers;
12. Volunteers with obvious gastrointestinal discomfort within 6 months before the start of the clinical trial;
13. Volunteers who have undergone gastrointestinal and liver surgery and those who have received any other surgery 6 months before the clinical trial;
14. The clinical laboratory examination is abnormal and the researchers judges that it has clinical significance;
15. Volunteers who have taken any clinical trial drugs within 3 months;
16. Volunteers who have used any antibiotics within 3 months;
17. Volunteers who have used any drug within 1 month;
18. Volunteers with hypertension （systolic blood pressure>139 mmHg，diastolic blood pressure>89 mmHg);
19. Volunteers with Parkinson's disease or family history of Parkinson's disease;
20. Volunteers with a family history of sudden cardiac death or arrhythmia;
21. Habitual drink, including coffee, tea, grapefruit juice and so on;
22. Significant weight loss recently;
23. Researcher judge that the volunteer has other factors that are not suitable for participating in this study, regardless of their severity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chinese volunteers who are planning to undergo gastrointestinal endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-10-31 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The activity and abundance of metabolism enzymes/transports in different section of gastrointestinal tract | Feb,2021-Sep, 2022
  LC-MS / MS will be used to quantitatively determine the activity of enzymes/transporters and protein content in mucosal samples including CYP1A2, CYP2C9, CYP2C19, CYP2D6, CYP2E1, CYP2J2, CYP3A4, CYP3A5, UGT1A1, UGT1A3, UGT1A4, UGT1A6, UGT1A7, UGT1A8, UGT1A10, UGT2B7, UGT2B17, ABCB1, ABCC2, ABCC3, ABCG2, ASBT, CNT1, CNT2, SGLT1, OATP2B1, OCTN1, OCIN2, OCT1, OCT3, PEPT1.
The physicochemical properties of gastric juice | Feb,2021-Sep, 2022
  The physicochemical properties of gastric juice including pH, viscosity, buffer capacity, osmotic pressure, and so on will be determined by means of pH-meter, rheometer, burette, freezing point depression, and so on
The composition of gastric juice | Feb,2021-Sep, 2022
  The composition of protein in gastric juice will be measured by LC-MS/MS or HPLC
The composition and content of bile acid in gastrointestinal mucosa, gastric juice and plasma | Feb,2021-Sep, 2022
  LC-MS/MS or HPLC will be used to determine the composition of bile acids in mucosal tissues, gastric juice and blood
The distribution of bacterial in gastrointestinal mucosa, saliva, gastric juice and feces | Feb,2021-Sep, 2022
  The distribution of bacteria in mucosa samples and gastric juice will be determined by high-throughput sequencing
The abundance of bacterial in gastrointestinal mucosa, saliva, gastric juice and feces | Feb,2021-Sep, 2022
  The abundance of bacteria in mucosa samples and gastric juice will be determined by high-throughput sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Dongyang Liu, Principal Investigator — Drug Clinical Trial Center
Locations (1):
- Dongyang Liu, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Den Abeele J, Rubbens J, Brouwers J, Augustijns P. The dynamic gastric environment and its impact on drug and formulation behaviour. Eur J Pharm Sci. 2017 Jan 1;96:207-231. doi: 10.1016/j.ejps.2016.08.060. Epub 2016 Sep 3. PMID 27597144
- [Background] Hayashi M, Matsumoto N, Takenoshita-Nakaya S, Takeba Y, Watanabe M, Kumai T, Takagi M, Tanaka M, Otsubo T, Kobayashi S. Individual metabolic capacity evaluation of cytochrome P450 2C19 by protein and activity in the small intestinal mucosa of Japanese pancreatoduodenectomy patients. Biol Pharm Bull. 2011;34(1):71-6. doi: 10.1248/bpb.34.71. PMID 21212520
- [Background] Berggren S, Gall C, Wollnitz N, Ekelund M, Karlbom U, Hoogstraate J, Schrenk D, Lennernas H. Gene and protein expression of P-glycoprotein, MRP1, MRP2, and CYP3A4 in the small and large human intestine. Mol Pharm. 2007 Mar-Apr;4(2):252-7. doi: 10.1021/mp0600687. Epub 2007 Jan 31. PMID 17263554
- [Background] Kalantzi L, Goumas K, Kalioras V, Abrahamsson B, Dressman JB, Reppas C. Characterization of the human upper gastrointestinal contents under conditions simulating bioavailability/bioequivalence studies. Pharm Res. 2006 Jan;23(1):165-76. doi: 10.1007/s11095-005-8476-1. Epub 2006 Dec 1. PMID 16308672
- [Background] Perez de la Cruz Moreno M, Oth M, Deferme S, Lammert F, Tack J, Dressman J, Augustijns P. Characterization of fasted-state human intestinal fluids collected from duodenum and jejunum. J Pharm Pharmacol. 2006 Aug;58(8):1079-89. doi: 10.1211/jpp.58.8.0009. PMID 16872555
- [Background] Vasapolli R, Schutte K, Schulz C, Vital M, Schomburg D, Pieper DH, Vilchez-Vargas R, Malfertheiner P. Analysis of Transcriptionally Active Bacteria Throughout the Gastrointestinal Tract of Healthy Individuals. Gastroenterology. 2019 Oct;157(4):1081-1092.e3. doi: 10.1053/j.gastro.2019.05.068. Epub 2019 Jun 5. PMID 31175864